CLINICAL TRIAL: NCT05497596
Title: The Association Between Human Microbiome and Vitamin D in Chronic Urticaria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH111-REC3-066
Record Dates: First submitted 2022-07-11; First posted 2022-08-11 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Urticaria
Keywords: Vitamin D; human microbiome; vitamin D receptors and vitamin D binding protein
MeSH Terms: conditions — Urticaria | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Vitamin D (2000IU/day) for 6 months
  Interventions: Other: Vitamin D
- Control group (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vitamin D — Vitamin D (2000IU/day) for 6 months
  Arms: Treatment group
Other: Placebo — Placebo
  Arms: Control group

SUMMARY:
A double-blind study to evaluate the role of human microbiome and vitamin D in the development of urticaria.

DETAILED DESCRIPTION:
Urticaria is a chronic allergic inflammatory disorder. Genetic and environmental factors, such as exposure to allergens and microbes, have a detrimental role in the development of chronic urticaria. Vitamin D also has an important role in urticaria. Lower sera vitamin D level was observed in patients that developed urticaria. Vitamin D binding protein (DBP) bound to vitamin D and regulated its metabolites in the circulation. Moreover, vitamin D receptors (VDR) have been identified on nearly all cells of the immune system. It may contribute to maintenance of intestinal barrier function by preventing increased intestinal permeability, dysbiosis, inflammation, and a lack of immune tolerance in the gut.

The investigators plan to design a double-blind trial to evaluate the role of human microbiome and vitamin D in the development of urticaria. We will enroll children with chronic urticaria (CU) and age and gender matched healthy children,and collected their venous blood and microbiome samples of nasal and anal swab. Then, CU subjects will be given vitamin D or placebo for 6 months in a randomized, double-blind way. After six months of follow-up, their blood, nasal cavity, and intestinal bacterial samples were taken. All microbial analysis, allergen detection, vitamin D concentration, VDR, DBP genotype will be analyzed by the core laboratory and bioinformatics center of CMUH.

The investigators believe this study can answer the cause-effect relationships of microbiota and vitamin D in the development of CU, and design a microbiota-related preventive and treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Experimental group: patients with chronic spontaneous urticaria under the age of 18 .
2. Control group: healthy children under the age of 18 (eg, healthy siblings of sick children).

Exclusion Criteria:

1. Recruit patients who have used antibiotics, systemic steroids, and immunosuppressants in the previous month.
2. Patients with C1 esterase inhibitor deficiency, lymphocytopenia, thrombocytopenia, severe diseases involving heart, liver, or kidney, metabolic disease, or autoimmune disease.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Levels of vitamin D | Month 0
  Vitamin D will be measured in a blood sample by ELISA to determine baseline status.
Levels of vitamin D | Month 6
  Vitamin D will be measured in a blood sample to follow the change from baseline in vitamin D level at month 6.
Single nucleotide polymorphism of vitamin D receptor and vitamin D binding protein. | Month 0
  Single nucleotide polymorphism (SNP) genotyping will be performed in a blood sample by using TaqMan SNP genotyping assays.
Microbiome Microbiome | Month 0
  Nasal and anal swabs will be used to detect respiratory and intestinal microbiome by using 16S rRNA sequencing to determine baseline status.
Microbiome Microbiome | Month 6
  Nasal and anal swabs will be used to detect respiratory and intestinal microbiome by using 16S rRNA sequencing,and to follow the change from baseline in microbiome at month 6.
Total IgE | Month 0
  Plasma total IgE concentration will be measured by microparticle immunoassay (IMx analyzer, Abbott Laboratories, Abbott Park, IL) and ELISA to determine baseline status.
Total IgE | Month 6
  Plasma total IgE concentration will be measured by microparticle immunoassay (IMx analyzer, Abbott Laboratories, Abbott Park, IL) and ELISA to follow the change from baseline in total IgE at month 6.
Allergen-specific IgE | Month 0
  Plasma allergen-specific IgE will be measured by BioIC ®.

SECONDARY OUTCOMES:
Quality of Life Assessment | Month 0 to Month 6
  Patients will rate their CU symptoms and the impact of their CU on various aspects of their lives. Each question is scored from 0 (not at all) to 3 (very much). Overall score, on scale of 0 to 57.
The Urticaria Activity Score 7 (UAS7) | Month 0 to Month 6
  The Urticaria Activity Score 7 measures number the weekly average of hives and pruritus measured twice a day. It scores from 0 to 42.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan